CLINICAL TRIAL: NCT02225106
Title: Dopamine Receptor Imaging to Predict Response to Stimulant Therapy in Chronic TBI
Acronym: DAPET-TBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140169; 14-N-0169
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Cognition Disorder; Attention Deficit Disorder; Traumatic Brain Injury
Keywords: Dopamine Receptors; Methylphenidate; Traumatic Brain Injury; C-11 Raclopride; Dopamine Release
MeSH Terms: conditions — Cognition Disorders; Attention Deficit Disorder with Hyperactivity; Brain Injuries, Traumatic | interventions — Methylphenidate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label methylphenidate treatment (Experimental): Forced titration with methylphenidate up to a dose of 30 mg administered orally twice daily.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Subjects will be treated with oral methylphenidate, using a forced titration up to a dose of 30 mg given twice daily for 4 weeks. At that point, the neuropsychologic tests are repeated.
  Other Names: Open label methylphenidate administration

SUMMARY:
Deficits in memory, attention, cognitive, and executive functions are the most common disabilities after traumatic brain injury (TBI). Dopamine (DA) neurotransmission is implicated in these neural functions and dopaminergic pathways are recognized to be frequently disrupted after TBI. Methylphenidate increases synaptic DA levels by binding to presynaptic dopamine transporters (DAT) and blocking re-uptake.

The objectives of this study are to use PET imaging with [11C]-raclopride, a D2/D3 receptor ligand, before and after administering methylphenidate, to measure endogenous DA release in patients who are experiencing problems with cognition, attention and executive function in the chronic stage after TBI. In addition, we will use TMS to test short intracortical inhibition, a gamma-aminobutyric acid receptor A (GABAA) - mediated phenomenon, which is under partial DA control, as a measure of dopaminergic activity on and off

DETAILED DESCRIPTION:
Deficits in memory, attention, cognitive, and executive functions are the most common disabilities after traumatic brain injury (TBI). Dopamine (DA) neurotransmission is implicated in these neural functions and dopaminergic pathways are recognized to be frequently disrupted after TBI. One of the most widely used DAergic drugs is methylphenidate (Ritalin ). Methylphenidate increases synaptic DA levels by binding to presynaptic dopamine transporters (DAT) and blocking re-uptake. PET with methylphenidate challenge to measure tonic DA release provides valuable insight into the molecular basis of attention-deficit hyperactivity disorder (ADHD) and addiction, as well as practical information regarding likely effectiveness of therapy (1). The objectives of this study are to use PET imaging with [11C]-raclopride, a D2/D3 receptor ligand, before and after administering methylphenidate, to measure endogenous DA release in patients who are experiencing problems with cognition, attention and executive function in the chronic stage after TBI. In addition, we will use TMS to test short intracortical inhibition, a gamma-aminobutyric acid receptor A (GABAA) - mediated phenomenon, which is under partial DA control, as a measure of dopaminergic activity on and off

methylphenidate.

STUDY POPULATION:

Males and females (n=30), between the ages of 18 and 55 years in the chronic stage after TBI who experience deficits in neuropsychological function from TBIs incurred 6 months after the injury, will be recruited from military treatment facilities or civilian clinics when presenting for clinical management of TBI or postconcussive symptoms.

DESIGN:

1. Study participants will be evaluated using brain MRI, psychometric measures adapted from the TBI Common Data Elements, attention tests and information about details of the injury and experience of post-concussive symptoms will be recorded. Transcranial magnetic stimulation (TMS) with placebo and with methylphenidate (60 mg by mouth) challenge will be performed to predict a stimulant response.
2. Subjects will be studied with [11C]-raclopride PET in two imaging sessions. One session will be after administration of placebo and the other after methylphenidate, 60 mg by mouth. Both placebo and methylphenidate will be given 60 minutes prior to injection of [11C]-raclopride to allow for peak uptake of methylphenidate in the brain. The binding potential of [11C]-raclopride relative to a non-displaceable reference region (cerebellum), BPND, will be used as a measure of D2/D3 receptor availability. The difference in BPND between methylphenidate and placebo ( BPND) is used to measure of tonic DA release.
3. Subjects will then be treated with oral methylphenidate, using a forced titration up to a dose of 30 mg given twice daily for 4 weeks. At that point, the neuropsychologic tests are repeated.

OUTCOME MEASURES:

The primary outcome is change in information processing speed

during neuropsychologic testing

ELIGIBILITY:
* INCLUSION:

To be included in the protocol, study participants must meet the following criteria:

1. Age 18 - 55 years, inclusive
2. A history of having sustained a moderate or severe TBI >= 6 months prior to enrollment. Evidence will be any one of the following 3 criteria:

   1. GCS 3 - 12 (GCS obtained in Emergency Room and noted in medical record)
   2. Post-traumatic amnesia > 24 hours
   3. TBI-related abnormality on neuroimaging (either CT or MRI). (Some missing information about the initial injury (i.e., documentation of initial GCS) is not necessarily exclusionary if the bulk of the available history indicates that the patient suffered a TBI and meets the inclusion criteria)
3. Persistent post-concussive symptoms, according to the DSM-IV Research Criteria for

   Post-Concussional Disorder, including:

   a) Difficulty in attention or memory. b) One or more of the following symptoms, which started shortly after the trauma and persist for at least three months: i) Fatigability ii) Disordered sleep iii) Changes in personality iv) Apathy or lack of spontaneity c) Symptoms in criteria (a) and (b) must have their onset after trauma, or there was a significant worsening of pre-existing symptoms after trauma.

   d) Disturbance from these symptoms causes significant impairment of social or occupational functioning and represents a significant decline from previous level of functioning.
4. Ability to read, write, and speak English
5. Ability to give informed consent.

EXCLUSION:

1. Evidence of penetrating brain injury.
2. Contraindication to methylphenidate therapy:

   1. Known glaucoma (consistently raised intraocular pressure with or without associated optic nerve damage)
   2. Motor tics or a family history of Tourette's syndrome (diagnosed by presence of both multiple motor and one or more vocal tics over the period of a year, with no more than three consecutive tic-free months)
   3. Known hypersensitivity to methylphenidate (hives, difficulty breathing, and swelling of face, lips, tongue, or throat).
   4. Known severe anxiety or restlessness which prevents from doing day to day activities.
   5. Known preexisting hypertension, heart failure, myocardial infarction, or ventricular arrhythmia.
   6. Known preexisting psychosis, bipolar illness.
   7. History of seizures, or interictal epileptiform discharges (IEDs) on EEG in absence of seizures.
   8. Known peripheral vasculopathy, including Raynaud s phenomenon.
   9. History of drug dependence or alcoholism.
   10. Concomitant treatment with coumadin anticoagulants, anticonvulsants (e.g., phenobarbital, phenytoin, primidone), and tricyclic drugs (e.g., imipramine,clomipramine, desipramine).
   11. Concomitant therapy with monoamine oxidase inhibitors (such as Marplan (isocarboxazid), Nardil (phenelzine), Emsam (selegiline), and Parnate (tranylcypromine)
   12. Concomitant treatment with blood pressure medication (both for high and low blood pressure).
   13. Pregnancy
   14. Breastfeeding
3. History or evidence of disabling pre-existing or co-existing disabling neurologic or psychiatric disorders not related to TBI, such as:

   1. Multiple sclerosis, pre- or co-existing
   2. Stroke (other than stroke at the time of TBI)
   3. Pre-existing disabling developmental disorder
   4. Pre-existing epilepsy
   5. Pre-existing major depressive disorder, aggressive behavior, hostility
   6. Pre-existing schizophrenia
4. Contraindication to MRI scanning

   1. Ferromagnetic metal in the cranial cavity or eye, e.g., aneurysm clip, implanted neural stimulator, cochlear implant, or ocular foreign body
   2. Implanted cardiac pacemaker or auto-defibrillator or pump
   3. Non-removable body piercing
   4. Claustrophobia
   5. Inability to lie supine for two hours
5. Contraindication to TMS, such as metal in the cranial cavity or implanted electronic hardware.
6. Current participation in other interventional clinical trial
7. Non-adherence to use of effective method of contraception for females of able to become pregnant for time from enrollment to the study until 2 weeks after completion of the study drug.
8. Present history of alcohol and substance abuse disorder determined (by DSM-IV).
9. Body mass index (BMI) > 40

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-N-0169.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Methylphenidate Treatment
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Methylphenidate Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 33 [24 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Maryland, United States
  participants
    United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Perceptual Organization and Processing Speed Index
Description: Relationship between tonic DA release (assessed by displacement of [11C] raclopride by oral methylphenidate) and improvement in processing speed after 4 weeks of treatment with oral methylphenidate.
  The Perceptual organization and processing speed index is measured from the Digit Symbol and Symbol Searches from the Weschler Adult Intelligence Scale (WAIS-IV). The tasks that comprise the PSI, (Coding, Symbol Search), are timed and require attending to visual material, visual perception and organization, visual scanning, and hand-eye coordination. It is a standardized scale were 100 is the mean of a normal population, and each 10 points represents 1 standard deviation above or below the mean. Thus, an index of 110 is 1 SD above the mean, 90 is 1 SD below the mean.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Methylphenidate Treatment
Number analyzed (Participants) | 11
score on a scale | 89 (10)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse events and serious adverse events were collected through structured questionnaires administered at the last study visit.
Arm/Group | Open Label Methylphenidate Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Methylphenidate Treatment (N=11)
Insomnia (Nervous system disorders) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02225106/Prot_SAP_ICF_000.pdf